CLINICAL TRIAL: NCT00005445
Title: Epidemiology of Pediatric Asthma Hospitalization
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4374; R29HL052076 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To study three possible, but yet unproven, influences on pediatric asthma hospitalization rates - diagnostic substitution, different systems of medical care, and asthma medication use.

DETAILED DESCRIPTION:
BACKGROUND:

Recent research has shown that asthma admission rates for children vary widely across geographic areas and have increased nationally for the past decade. The results from these studies will have direct relevance to the clinical care and development of public policy for children with asthma.

DESIGN NARRATIVE:

Specific hypotheses regarding these factors which influence pediatric asthma hospitalization were tested in two different data sets: ecologic studies of trends and area variations of the children residing in the contiguous states of Maine, New Hampshire, and Vermont for 1980 - 1994; retrospective cohort analyses of children enrolled at a staff model HMO, Group Health Cooperative of Puget Sound for 1977 - 1994. These studies utilized detailed information regarding area and individual 'exposure' to differing systems of health care and asthma medications, controlling for socioeconomic status.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-04; Study Completion 1999-02

REFERENCES:
- [Background] Goodman DC, Fisher E, Stukel TA, Chang C. The distance to community medical care and the likelihood of hospitalization: is closer always better? Am J Public Health. 1997 Jul;87(7):1144-50. doi: 10.2105/ajph.87.7.1144. PMID 9240104
- [Background] Goodman DC, Littenberg B, O'Connor GT, Brooks JG. Theophylline in acute childhood asthma: a meta-analysis of its efficacy. Pediatr Pulmonol. 1996 Apr;21(4):211-8. doi: 10.1002/(SICI)1099-0496(199604)21:43.0.CO;2-R. PMID 9121849
- [Background] Goodman DC, Lozano P, Stukel TA, Chang Ch, Hecht J. Has asthma medication use in children become more frequent, more appropriate, or both? Pediatrics. 1999 Aug;104(2 Pt 1):187-94. doi: 10.1542/peds.104.2.187. PMID 10428993
- [Background] Goodman DC, Stukel TA, Chang CH. Trends in pediatric asthma hospitalization rates: regional and socioeconomic differences. Pediatrics. 1998 Feb;101(2):208-13. doi: 10.1542/peds.101.2.208. PMID 9445493
- [Background] Goodman DC, Fisher ES, Bubolz TA, Mohr JE, Poage JF, Wennberg JE. Benchmarking the US physician workforce. An alternative to needs-based or demand-based planning. JAMA. 1996 Dec 11;276(22):1811-7. doi: 10.1001/jama.276.22.1811. PMID 8946901